CLINICAL TRIAL: NCT04675658
Title: Stay Active Physical Activity Program for Teachers, Students, and Families
Brief Title: Stay Active Physical Activity Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00001495
Record Dates: First submitted 2020-12-08; First posted 2020-12-19 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Healthy Lifestyle; Sedentary Behavior
Keywords: Physical Activity; Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care provider/study staff will be masked to the arm the participant is assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Classroom Intervention (Active Comparator): Physical activity support is provided by integrating daily structured activities in the classroom delivered by physical activity leaders through a video conferencing platform in partnership with the classroom teacher. Activities last about 10 minutes or less and have the flexibility of being integrated with academic lessons or serving as a break from academics.
  The activities are simple and get kids moving in place. The activities will be delivered by a research staff member via video conferencing (using the schools preferred platform). A combination of live activities led by the research team and pre-recorded videos will be used (see example below). If live videos do not work for the teacher, they will have the option to only use the pre-recorded videos or receive a list of resources to promote CBPA in their classrooms.
  Interventions: Behavioral: CBPA
- Classroom Intervention plus family support (Experimental): Same components as the Classroom Intervention Arm plus the following:
  Family Component: A newsletter will be sent to parents or guardians once every two weeks over the semester and posted on the study website. The newsletters include physical activity information related to safety/protection, skills building, motivation, overcoming barriers, and goal setting and monitoring (all newsletters are included as an appendix). As part of the program, children also receive a Garmin wearable physical activity monitor. Parents or guardians will receive text messages with behavior change messages based on the Garmin data (text message content is included as an appendix). Text messages also contain links to website materials.
  Texts will be sent out using the Twilio platform.
  Interventions: Behavioral: CBPA + family support

INTERVENTIONS:
Behavioral: CBPA + family support — Classroom Based Physical Activity + family support as described in the Arm
  Arms: Classroom Intervention plus family support
Behavioral: CBPA — Classroom Based Physical Activity
  Arms: Classroom Intervention

SUMMARY:
The pilot study will create, implement, and evaluate a physical activity program in both the school and home setting during the COVID-19 pandemic.

DETAILED DESCRIPTION:
This study will compare the impact of two physical activity interventions on student's physical activity.

ELIGIBILITY:
Inclusion Criteria:

Classrooms

* Teacher of a 4th or 5th grade class in the Kansas City area.
* English speaking only

Students

* Any student in the selected classrooms
* A parent or guardian of the student
* English speaking only

Exclusion Criteria:

* Does not meet the required criteria above.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-10-05 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Daily minutes of PA (physical activity) | 3 months
  Measured by Garmin device
Daily step count | 3 months
  Measured by Garmin device

SECONDARY OUTCOMES:
Parent perceptions of interventions | 3 months
  Measured via satisfaction surveys
Teacher perceptions of interventions | 3 months
  Measured via satisfaction interviews

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Carlson, PhD, Principal Investigator — Research Faculty
Locations (1):
- Children's Mercy, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04675658/Prot_SAP_000.pdf